CLINICAL TRIAL: NCT04582955
Title: Chidamide Combined With Neoadjuvant Chemotherapy in Early Triple-negative Breast Cancer
Brief Title: Neoadjuvant Treatment of Early Triple-negative Breast Cancer With Chidamide and Chemotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSIIT-C03
Record Dates: First submitted 2020-09-28; First posted 2020-10-12 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2020-11

CONDITIONS: Triple-negative Breast Cancer
Keywords: neoadjuvant; Chidamide; triple-negative breast cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm A (Experimental): Chidamide, orally,20mg at day 0,4,7,11,21,every 3 weeks; in combination with Docetaxel 75mg/m2,intravenous infusion，at day1 every 3 weeks，and Epirubicin 75mg/m2, intravenous infusion，at day1 every 3 weeks
  Interventions: Drug: Chidamide in combination with chemotherapy

INTERVENTIONS:
Drug: Chidamide in combination with chemotherapy — Chidamide, orally,20mg at day 0,4,7,11,21,every 3 weeks; in combination with Docetaxel 75mg/m2,intravenous infusion，at day1 every 3 weeks，and Epirubicin 75mg/m2, intravenous infusion，at day1 every 3 weeks
  Other Names: Other Name: For Chidamide: HBI-8000, CS055

SUMMARY:
Objective to evaluate the efficacy and safety of neoadjuvant therapy with Chidamide combined with chemotherapy for stage II - III triple-negative breast cancer，and to compare the efficacy and safety of chemotherapy with Chidamide and chemotherapy alone in the neoadjuvant treatment of stage II - III triple-negative breast cancer

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤ 70, postmenopausal / premenopausal women;
2. Patients with unilateral or bilateral primary invasive triple-negative (ER expression < 1%, PR < 1%, and HER2 negative *) confirmed by histology or cytology;
3. non-metastatic invasive TNBC（stage II-III）with at least one axillary lymph node involvement (T1cN1-2M0 or T2-3N1-2M0);
4. previously untreated for breast cancer;
5. There was at least one measurable primary lesion (according to RECIST v1.1);
6. ECoG score 0-1;
7. Adequate organ and marrow function as defined below:

   absolute value of neutrophils ≥ 1.5 × 109 / L, platelets ≥ 100 × 109 / L, hemoglobin≥ 90 g / L;
8. Volunteer to participate in this clinical trial and sign written informed consent

Exclusion Criteria:

1. No measurable lesions, such as pleural or pericardial effusion, ascites, etc;
2. Major surgical procedures or significant trauma were performed within 4 weeks before enrollment, or patients were expected to receive major surgical treatment (not related to breast cancer);
3. Previously treated with chemotherapy or HDAC inhibitors (including romidepsin, vorinostat, belinostat, and panobinostat，etc);
4. Have allergic history to the components of this regimen;
5. Treated with radiotherapy within 4 weeks before admission;
6. Have a history of immunodeficiency, including HIV positive, or other acquired or congenital immunodeficiency diseases, or have a history of organ transplantation;
7. Uncontrolled cardiovascular diseases, history of clinically significant QT interval prolongation, or QTc interval > 450 ms at screening;
8. Abnormal liver function [total bilirubin > 1.5 times of the upper limit of normal value; ALT / AST > 2.5 times of upper limit of normal value for patients without liver metastasis ; ALT / AST > 5 times of upper limit of normal value for patients with liver metastasis ], abnormal renal function (serum creatinine > 1.5 times of upper limit of normal value);
9. Pregnant, lactating or fertile women with a positive baseline pregnancy test; or subjects of childbearing age who are not willing to take effective contraceptive measures during the study period and at least 8 weeks after the last administration;
10. According to the judgment of the investigator, there are some concomitant diseases (such as severe hypertension, diabetes, thyroid disease, active infection, etc.) that seriously endanger the safety of patients or affect patients to complete the study;
11. A clear history of epilepsy or dementia, including neurological disorders;
12. The investigator determined not suitable to participate in this study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Enrollment: 20 (Estimated)
Dates: Start 2020-10-30 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy Outcome: pathologic complete response（pCR） rate（ypT0/is ypN0） | 1years
  pCR defined as no invasive tumour residuals in breast and no invasive and no non-invasive tumour residuals in axillary lymph nodes (ypT0/is ypN0) after neoadjuvant therapy

SECONDARY OUTCOMES:
Objective Response Rate (ORR) by RECIST v1.1 | 12 months
  Objective Response Rate (ORR) by RECIST v1.1
pCR by other definitions | 12 months
  response by other pCR definitions（ypT0 ypN0; ypT0 ypN0/+;ypT0/is ypN0/+; ypT[any] ypN0）
Breast conserving surgery rate | 12 months
  Breast conserving surgery rate
Event-free survival | 60 months
  Event-free survival
Overall survival | 72 months
  Overall survival
Incidence of Adverse Events (AEs) | 12 months
  Incidence of Adverse Events (AEs)

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Hospital, Tianjin, Tianjin Municipality, China